CLINICAL TRIAL: NCT07078955
Title: A Phase 2, Multicenter, Randomized, Open-Labeled, Artificial Tear-Controlled, 6-Week Clinical Study to Assess the Dose Regimen, Safety and Efficacy of BRM421 Ophthalmic Solution in Patients With Dry Eye Disease
Brief Title: A Dose Regimen Study of BRM421 Ophthalmic Solution in Patients With Dry Eye Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BRIM Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRM421-24-C001
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Dry Eye Disease (DED); Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Lubricant Eye Drops

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Artificial Tear (Other)
  Interventions: Drug: Artificial Tear
- BRM421 Ophthalmic Solution, 0.03% (Active Comparator)
  Interventions: Drug: BRM421 Ophthalmic Solution, 0.03%
- BRM421 Ophthalmic Solution, 0.06% (Active Comparator)
  Interventions: Drug: BRM421 Ophthalmic Solution, 0.06%

INTERVENTIONS:
Drug: BRM421 Ophthalmic Solution, 0.03% — A topical drop of 0.03% BRM421 ophthalmic solution.
  Arms: BRM421 Ophthalmic Solution, 0.03%
Drug: Artificial Tear — A topical drop of Artificial Tear.
  Arms: Artificial Tear
Drug: BRM421 Ophthalmic Solution, 0.06% — A topical drop of 0.06% BRM421 ophthalmic solution.
  Arms: BRM421 Ophthalmic Solution, 0.06%

SUMMARY:
To evaluate the safety and efficacy of BRM421 Ophthalmic Solution compared to artificial tear for treatment of the signs and symptoms of dry eye disease (DED)

ELIGIBILITY:
Inclusion Criteria:

* Are ≥18 years of age;
* Are willing and able to comply with all study procedures and restrictions and the visit schedule;
* Have a self-reported history of dry eye prior to enrollment;
* If a woman of childbearing potential (WOCBP): are non-lactating, have a negative urine pregnancy test (UPT), and agree to use an acceptable form of contraception for the duration of the study;

Exclusion Criteria:

* Within 3 months prior to Visit 1, have participated in any other investigational study or used an investigational product or device;
* Have any history of organ or bone marrow transplant, immunodeficiency disorder, human immunodeficiency virus, or hepatitis C, or any evidence of acute active hepatitis A (anti-hepatitis A virus immunoglobulin M);
* Have any significant illness or condition that, in the opinion of the Investigator, could affect the study outcome measures. Such illnesses include (but are not limited to) Sjögren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, severe cardiopulmonary disease, poorly controlled hypertension or diabetes, or drug/alcohol addiction;
* Within 12 months prior to Visit 1, have undergone any ocular surgical procedure, including laser-assisted in situ keratomileusis (LASIK) or a similar corneal refractive surgery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total corneal fluorescein staining (tCFS) score | 6 weeks
  Total corneal fluorescein staining (tCFS) score by using NEI Scale (0-20, higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- New Taipei Municipal TuCheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No